CLINICAL TRIAL: NCT03779100
Title: Lenvatinib Plus Programmed Cell Death Protein-1 (PD-1) Antibody for Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Lenvatinib Plus PD-1 Antibody for Unresectable ICC
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol modification
Sponsor: Shi Ming (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S075
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; Lenvatinib; PD-1 Antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib Plus PD-1 (Experimental): Participants received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the participant's body weight less than (<) 60 kg at baseline, orally, once daily (QD) in continuous 14-day treatment cycles, and received 3mg/kg PD-1 antibody intravenously every 2 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Lenvatinib; Drug: PD-1 antibody

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
  Other Names: E7080, Lenvima
Drug: PD-1 antibody — 3mg/kg intravenously every 2 weeks
  Other Names: Programmed cell death 1 antibody

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib combined with PD-1 antibody for patients with unresectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ICC
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* Chemotherapy resistance or patient refuse chemotherapy
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* Without distant metastasis, but intrahepatic lymph node metastasis is allowed
* The following laboratory parameters:

Platelet count ≥ 50,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China